CLINICAL TRIAL: NCT04443296
Title: Study of Tumor Infiltrating Lymphocytes Following Concurrent Chemoradiotherapy in the Treatment of Patients With Cervical Carcinoma
Brief Title: Study of Tumor Infiltrating Lymphocytes Following CCRT in the Treatment of Patients With Cervical Carcinoma
Acronym: TIL-Cx
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jihong Liu, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYSGO008
Record Dates: First submitted 2020-06-20; First posted 2020-06-23 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Cervical Carcinoma
Keywords: Tumor Infiltrating Lymphocytes; Concurrent chemotherapy
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CCRT+TIL (Experimental): Cisplatin based concurrent chemoradiotherapy(CCRT) combined with tumor-infiltrating lymphocyte (TIL)
  Interventions: Drug: CCRT+TIL

INTERVENTIONS:
Drug: CCRT+TIL — Cisplatin based chemotherapy concurrently with radiotherapy, then TIL infusing following concurrent chemoradiotherapy

SUMMARY:
A Phase I trial to evaluate the feasibility, toxicity and effectiveness of cisplatin concurrent chemoradiotherapy plus TIL in treating patients with FIGO stage IIIA to IVA cervical carcinoma.

DETAILED DESCRIPTION:
Concurrent chemoradiotherapy (CCRT) was the standard treatment for locoregionally advanced cervical cancer, while the incidence of treatment failure is still high. Adjuvant chemotherapy or inducing chemotherapy addition to CCRT did not significantly improve patient survival compared to CCRT alone. Hence, there is a need for novel therapies to improve survival for these patients.

Accumulating evidence shows that tumor-infiltrating lymphocytes (TILs) selected for tumor recognition and greatly expanded in vitro are effective for treating cervical cancer patients.

This is a phase I trial to evaluate the feasibility, toxicity and effectiveness of cisplatin concurrent chemoradiotherapy plus TIL in treating patients with FIGO stage IIIA to IVA cervical carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically proven squamous cell carcinoma, adenocarcinoma or adenosquamous carcinoma of the cervical uteri
* Patients with stage IIIA-IVA cervical cancer according to the International Federation of Gynecology and Obstetrics (FIGO)
* Patients who were ≥ 18 and ≤ 70 years old
* Patients with an ECOG performance status of 0, 1, or 2
* Adequate hematological, renal, and hepatic functions defined as:

granulocytes ≥ 1.5 x 109/L, platelets ≥ 100 x 109/L, total bilirubin, ALT and AST ≤ 1.5 x upper normal limit, creatinine ≤ upper normal limit

* Patients provided written, voluntary informed consent
* Patients who were accessible to follow up and management in the treatment center

Exclusion Criteria:

* Patients with past or current history of malignancy other than the entry diagnosis except for a "cured" malignancy more than five years prior to enrollment
* Patients who received previous chemotherapy or radiotherapy
* Patients with active angina or documented myocardial infarction within the 6 months preceding registration and patients with a history of significant ventricular arrhythmia requiring medication or congestive heart failure, as well as a history of 2nd or 3rd degree heart blocks
* Patients with an active infection or other serious underlying medical conditions that would impair the ability of the patient to receive the planned treatment, including prior allergic reactions to drugs containing platinum
* Patients with dementia or altered mental status that would prohibit the understanding and providing of informed consent
* Patients with inadequate caloric and/or fluid intake

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-10-12 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Toxicity Evaluation | From chemo-radiotherapy start until Day30 after TIL infusion
  Patients will be monitored for clinical toxicity by by the National Cancer Institute Common Terminology Criteria for Adverse Events.
Feasibility of CCRT in combination with TIL successful infusion | 30 days after start of TIL-ACT infusion
  Number of patients receiving a complete TIL infusion

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 1, 3, 6, 9, 12 months
  Disease response evaluated after the completion of the chemoradiotherapy and TIL treatment. Achievement of complete response, partial response.
Disease control rate (DCR) | 1, 3, 6, 9, 12 months
  Disease response evaluated after the completion of the chemoradiotherapy and TIL treatment. Achievement of complete response, partial response or stable disease.
Disease control time (DCT) | 1, 3, 6, 9, 12 months
  Duration from complete response, partial response or stable disease to progression.
Immunological correlates to tumor response | 1, 3, 6, 9, 12 months
  Post-hoc exploratory analyses for immunological correlates to tumor response.

CONTACTS AND LOCATIONS:
Overall Officials: Jihong Liu, MD, Study Director — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huang H, Nie CP, Liu XF, Song B, Yue JH, Xu JX, He J, Li K, Feng YL, Wan T, Zheng M, Zhang YN, Ye WJ, Li JD, Li YF, Li JY, Cao XP, Liu ZM, Zhang XS, Liu Q, Zhang X, Liu JH, Li J. Phase I study of adjuvant immunotherapy with autologous tumor-infiltrating lymphocytes in locally advanced cervical cancer. J Clin Invest. 2022 Aug 1;132(15):e157726. doi: 10.1172/JCI157726. PMID 35727633